CLINICAL TRIAL: NCT01495104
Title: A SINGLE CENTER, OPEN LABEL, FIXED SEQUENCE, TWO-PERIOD STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSE VALPROATE ON THE PHARMACOKINETICS OF RO4917838 AND VICE VERSA IN HEALTHY MALE VOLUNTEERS
Brief Title: A Study on the Effects of Valproate on the Pharmacokinetics of RO4917838 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25258; 2011-002256-14 (EudraCT Number)
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Valproic Acid

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO4917838; Drug: valproate

INTERVENTIONS:
Drug: RO4917838 — Multiple doses
Drug: valproate — Multiple doses

SUMMARY:
This open-label, fixed-sequence, two-period study will assess the effect of multiple dose valproate on the pharmacokinetics of RO4917838 at steady state and vice versa in healthy male volunteers. In Period 1, subjects will receive valproate for 5 days. After a washout period of 5 days to 2 weeks, subjects will receive, in Period 2, RO4917838 for 15 days with concomitant valproate on Days 11-15. Anticipated time on study is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18 to 65 years of age inclusive
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Healthy as determined by the investigator on the basis of medical/surgical history, physical examination, clinical laboratory test results, vital signs, and a 12-lead electrocardiogram (ECG)
* Non smoker or smoker of fewer than 10 cigarettes per day

Exclusion Criteria:

* History of alcoholism, drug abuse or addiction within the last year prior to Day -1 of the study
* Alcohol consumption averaging more than 24 g of alcohol per day
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, psychiatric disease, or cancer
* Any major illness within the 4 weeks prior to dosing or any acute disease state (e.g. nausea, vomiting, fever, diarrhea) within 7 days of study Day -1
* Any confirmed allergic reactions against any drug, or multiple allergies in the judgment of the investigator
* Positive for hepatitis B, hepatitis C or HIV infection
* Involvement in other investigational studies of any type within 90 days of first study drug administration or within 5 times the elimination half-life of the tested drug, whichever is longer

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effect of valproate multiple-dose administration on pharmacokinetics of RO4917838 at steady-state: Area under the concentration-time curve (AUC) | Period 2, day 10 and day 15
Effect of RO4917838 multiple-dose administration on the pharmacokinetics of valproate at steady state: Area under the concentration-time curve (AUC) | Period 1, day 5 and Period 2, Day 15

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rueil-Malmaison, France